CLINICAL TRIAL: NCT06167109
Title: Endoscopic NBI Combined With MRI to Guide the Optimization of Clinical Target Volume Delineation in Eccentric Nasopharyngeal Carcinoma
Brief Title: NBI Combined With MRI to Guide CTV Optimization in Eccentric Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Wang, Associate Director of Chongqing University Cancer Hospital, Chongqing University Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPC-CTV
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Nasopharyngeal Carcinoma by AJCC V8 Stage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimized CTV (Experimental): The contralateral CTV1 was defined as a subclinical disease consisting of 5mm margin surrounding GTVnx.The CTV2 was defined as potentially involved regions consisting of 5mm margin surrounding CTV1, and contralateral CTV2 only included the pharyngeal recess.
  Interventions: Radiation: CTV optimized IMRT
- Conventional CTV (No Intervention): The CTV1 was defined as GTVnx + 5 mm + entire nasopharynx mucosa .The CTV2 was defined as GTV1+ 5 mm + corresponding anatomical structures.

INTERVENTIONS:
Radiation: CTV optimized IMRT — The contralateral CTV1 was defined as a subclinical disease consisting of 5mm margin surrounding GTVnx.The CTV2 was defined as a potentially involved regions consisting of 5mm margin surrounding CTV1, and contralateral CTV2 only included the pharyngeal recess.
  Arms: Optimized CTV

SUMMARY:
This is a prospective, single-center clinical trial in eccentric nasopharyngeal carcinoma (NPC) patients. The aim of this study is to evaluate the efficacy and safety of NBI combined with MRI-guided optimized CTV compared with conventional CTV, and to compare the radiotherapy-related adverse events and quality of life between the two groups.

DETAILED DESCRIPTION:
All patients with eccentric nasopharyngeal carcinoma were selected on the basis of MRI findings and NBI endoscopy was performed in these patients. The patients were enrolled if both NBI endoscopy and MRI showed eccentric NPC. Patients with contralateral tissue mucosal abnormalities detected by NBI and confirmed by biopsy were excluded. Then the patients were randomly divided into an experimental group (Optimized CTV) or a control group (Conventional CTV) to evaluate the efficacy and safety of the two groups, as well as radiotherapy-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age;
2. ECOG Performance Status 0,1 or 2;
3. Pathologically diagnosed as nasopharyngeal carcinoma;
4. Pretreatment nasopharynx and neck MRI imaging;
5. Nasopharyngeal suspected lesions were examined by NBI endoscopy;
6. Meeting the definition of eccentric NPC with ipsilateral (affected side) staging of T1-4 and contralateral (healthy side) staging of T0;
7. Patients evaluated without contraindications to radiotherapy;
8. Voluntary participation in clinical research, and signed informed consent.

Exclusion Criteria:

1. Patients who did not successfully undergo all three examinations (MRI, NBI, and endoscopic biopsy);
2. Other rare pathological types, such as adenocarcinoma;
3. Patients with tumor invasion of the clivus;
4. Patients whose contralateral retropharyngeal lymph nodes met the diagnostic criteria;
5. Invasion of paranasal sinuses (except simple sphenoid invasion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Acute adverse reactions | 3 months
  The acute adverse reactions of patients during or after radiotherapy were evaluated with the corresponding standard scales.
Control rate of non-irradiated area | 36 months

SECONDARY OUTCOMES:
Local recurrence-free survival(LRFS) | 36 months
  The duration of time to LRFS was calculated from the date of histological diagnosis until documented treatment local failure or death from any cause.
Progress-free survival(PFS) | 36 months
  Defined as time from randomization to locoregional or distant metastasis relapse or death from any cause, whichever occurred first.
Overall survival (OS) | 36 months
  Overall survival is measured from day of diagnosis until death due to any cause or the latest known date alive.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, Ph.D, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Song Y, Wang Y, Yang M, Yu X, Li M, Long B, Shu X, Zhang X, Wang F, Wang C, Hu M, Sui JD, Wang Y. Individualization of clinical target volume delineation in eccentric nasopharyngeal carcinoma: a prospective comparative study. Front Oncol. 2025 Aug 4;15:1587764. doi: 10.3389/fonc.2025.1587764. eCollection 2025. PMID 40831921